CLINICAL TRIAL: NCT00885261
Title: The Prevalence of Metabolic Syndrome in Patients Suffering From Chronic Pain
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Silviu Brill MD, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-09-SB-096-CTIL
Record Dates: First submitted 2009-04-19; First posted 2009-04-21 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2009-04

CONDITIONS: Pain and Metabolic Syndrome
Keywords: chronic pain and metabolic syndrome
MeSH Terms: conditions — Pain; Metabolic Syndrome; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Obesity is considered as the epidemic of the century. Central obesity is one of the metabolic syndrome's features. It has been proven that obesity can cause back pain and headaches; thus, there might be a link between chronic pain and the syndrome.

The objective of this study is to assess the prevalence of metabolic syndrome in patients suffering from chronic pain.

DETAILED DESCRIPTION:
All patients will answer a questionnaire, their hip circumference will be measured, and their BMI will be calculated (weight/(height)2 ).

The patients' blood pressure will be measured. The patients will be asked to bring their blood tests (lipids and glucose).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 that suffer from chronic pain and are being treated at the pain medicine unit

Exclusion Criteria:

* Pregnant women, patients with abdominal wall defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 that suffer from chronic pain and are being treated at the pain medicine unit
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-05; Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silviu Brill, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Pain Medicine Unit, Tel Aviv, Israel